CLINICAL TRIAL: NCT03185299
Title: Impact of Reinforced Education by Video on the Quality of Bowel Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director, Head of Department of Gastroenterology, Principal Investigator, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIDEO
Record Dates: First submitted 2017-04-26; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Bowel Preparation Scale; Adenoma Detection Rate
Keywords: Polyp detection rate; Adenoma detection rate; Boston Bowel Preparation Scale
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): Patients randomized to the intervention arm will be contacted 48-72h before their procedure via telephone using a standardized script and will be provided a link to a website allowing posting of videos for public viewing
  Interventions: Other: Video
- Standard preparation instructions (Experimental): The control arm will receive written instruction on preparing for a colonoscopy per standard of care
  Interventions: Other: Standard preparation instructions

INTERVENTIONS:
Other: Video — Patients randomized to the intervention arm will be contacted 48-72h before their procedure via telephone using a standardized script and will be provided a link to a website allowing posting of videos for public viewing
  Arms: Video
Other: Standard preparation instructions — The control arm will receive written instruction on preparing for a colonoscopy per standard of care
  Arms: Standard preparation instructions

SUMMARY:
High quality bowel preparation is essential for successful colonoscopy. This study aimed to assess the impact of reinforced education by Video on the quality of bowel preparation. This prospective, endoscopist-blinded, randomized, controlled study was conducted. Reinforced education groups received additional education via reminders by video 2 days before colonoscopy. The primary outcome was the quality of the bowel preparation according to the Boston Bowel Preparation Scale (BBPS). The secondary outcomes included polyp detection rate (PDR), adenoma detection rate (ADR), tolerance, and subjective feelings of patients.

ELIGIBILITY:
Inclusion Criteria:

* outpatients aged 18-80 years
* referred for routine diagnostic colonoscopy
* with access to the educational video themselves or through close family members living in the same household were eligible.

Exclusion Criteria:

1. pregnancy or breastfeeding
2. allergy to purgatives
3. suspected intestinal obstruction, stricture, or perforation
4. hemodynamic instability
5. impaired swallowing reflex or mental status
6. severely medical status, such as New York Heart Association grade III or grade IV congestive heart failure and severe renal failure
7. illiteracy
8. history of oesophagus、stomach 、duodenum、small intestine or colorectal surgery
9. participation declined.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-07-04 (Estimated); Primary Completion 2018-06-04 (Estimated); Study Completion 2018-08-04 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | 2 days
  The primary end point of the study was adequate bowel prepara- tion quality de ned as a BBPS total score of ≥6 with all segment scores ≥2

SECONDARY OUTCOMES:
Polyp detection rate | 2 days
  Secondary end points included polyp detection rate which would be higher in the colonoscopy with satisfactory bowel preparation.
Adenoma detection rate | 2 days
  Secondary end points included adenoma detection rate which would be higher in the colonoscopy with satisfactory bowel preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Yu, Prof, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rice SC, Higginbotham T, Dean MJ, Slaughter JC, Yachimski PS, Obstein KL. Video on Diet Before Outpatient Colonoscopy Does Not Improve Quality of Bowel Preparation: A Prospective, Randomized, Controlled Trial. Am J Gastroenterol. 2016 Nov;111(11):1564-1571. doi: 10.1038/ajg.2016.450. Epub 2016 Oct 18. PMID 27753434